CLINICAL TRIAL: NCT05877053
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Multi-part, Single and Multiple Ascending Dose Study of CK-4021586 in Healthy Adult Participants
Brief Title: A Single and Multiple Ascending Dose Study of CK-4021586 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CY 9011
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: CK-586; CK-4021586

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- CK-4021586 for SAD Cohort (Experimental): Subjects will be assigned to one of 8 planned dose cohorts and receive single doses of CK-4021586
  Interventions: Drug: CK-4021586
- Placebo for SAD Cohort (Placebo Comparator): Subjects will be assigned to one of approximately 8 planned cohorts and receive single doses of placebo
  Interventions: Drug: Placebo for CK-4021586
- CK-4021586 for MAD Cohort (Experimental): Subjects will be assigned to one of 4 planned dose cohorts and receive multiple doses of CK-4021586
  Interventions: Drug: CK-4021586
- Placebo for MAD Cohort (Placebo Comparator): Subjects will be assigned to one of approximately 4 planned cohorts and receive multiple of placebo
  Interventions: Drug: Placebo for CK-4021586
- Food Effect (Experimental): Healthy subjects will be administered CK-4021586 with and without food in a cross-over fashion
  Interventions: Drug: CK-4021586

INTERVENTIONS:
Drug: CK-4021586 — CK-4021586
  Arms: CK-4021586 for MAD Cohort; CK-4021586 for SAD Cohort; Food Effect
Drug: Placebo for CK-4021586 — Placebo for CK-4021586
  Arms: Placebo for MAD Cohort; Placebo for SAD Cohort

SUMMARY:
The purposes of this study are to:

* Learn about the safety and tolerability of CK 4021586 after a single dose and multiple doses in healthy subjects.
* Find out how much CK-4021586 is in the blood after a single dose and multiple doses.
* Determine the effect different doses of CK-4021586 on the pumping function of the heart.
* Determine the effect of food in the stomach on how much CK-4021586 is in the blood after a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged between 18 and 55 years (inclusive) with a body mass index between 18.0 and 30.0 kg/m2 (inclusive), with a body weight > 50.0 kg

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic/immunologic, dermatologic, hepatic, renal, hematologic, respiratory, cardiovascular (including arrhythmia), gastrointestinal, gallbladder/biliary, musculoskeletal, neurologic, or psychiatric disorder in the opinion of the Investigator or designee.
* History of significant hypersensitivity or allergy to any drug compound or other substance, unless approved by the Investigator and the Sponsor's Medical Monitor.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, hernia repair, and/or cholecystectomy will be allowed).
* Participants with breast implants that may impede echocardiography
* Clinically significant illness within 4 weeks prior to check in.
* Significant ECG abnormalities (heart block, prolonged QT interval, arrhythmia)
* History of, or current substance abuse (drug or alcohol), known drug or alcohol dependence within the last 2 years prior to Screening, or positive test for drugs of abuse during the screening period
* Any acute or chronic condition that would limit the participant's ability to complete and/or participate in this clinical study, in the judgment of the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs | Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14; Time Frame for Food Effect Cohorts: Days 1 to 7 (Treatment Periods 1 and 2)
  To assess the safety and tolerability of CK-4021586 when administered orally as single or multiple doses to healthy participants

SECONDARY OUTCOMES:
Primary PK parameters of CK-4021586 including AUC | Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14; Time Frame for Food Effect Cohorts: Days 1 to 7 (Treatment Periods 1 and 2)
  To characterize the PK of CK-4021586 and CK-4022235 after single and multiple oral doses in healthy participants
Changes over time from baseline in echocardiographic parameters including, but not limited to, LVEF | Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14
  To characterize the PD effects of single and multiple oral doses of CK-4021586 in healthy participants

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Leadership at Cytokinetics, Study Director — Cytokinetics
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No